CLINICAL TRIAL: NCT03470545
Title: A Randomized, Double Blind, Placebo Controlled Clinical Study to Evaluate Mavacamten (MYK-461) in Adults With Symptomatic Obstructive Hypertrophic Cardiomyopathy
Brief Title: Clinical Study to Evaluate Mavacamten (MYK-461) in Adults With Symptomatic Obstructive Hypertrophic Cardiomyopathy
Acronym: EXPLORER-HCM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: MyoKardia, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MYK-461-005
Record Dates: First submitted 2018-03-12; First posted 2018-03-20 (Actual); Results first posted 2021-10-04 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2020-05

CONDITIONS: Obstructive Hypertrophic Cardiomyopathy
Keywords: Symptomatic, left ventricular outflow tract gradient
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — MYK-461

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- mavacamten (MYK-461) (Experimental)
  Interventions: Drug: mavacamten
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: mavacamten — mavacamten capsules
  Other Names: MYK-461
  Arms: mavacamten (MYK-461)
Drug: Placebo — placebo oral capsule
  Arms: Placebo

SUMMARY:
This is a multicenter, international, double-blind study of the administration of mavacamten in participants with symptomatic obstructive HCM (oHCM). Approximately 220 participants will be randomized to receive placebo or mavacamten.

ELIGIBILITY:
Key Inclusion Criteria:

* Age 18 and greater, body weight ≥ 45kg
* Has adequate acoustic windows to enable accurate transthoracic echocardiograms (TTEs)
* Diagnosed with oHCM consistent with current American College of Cardiology Foundation/American Heart Association and European Society of Cardiology guidelines and satisfy both criteria:
* Has documented left ventricular ejection fraction (LVEF) ≥55%
* NYHA Class II or III
* Has documented oxygen saturation at rest ≥90% at Screening
* Is able to perform an upright CPET and has a respiratory exchange ratio (RER) ≥1.0 at Screening per central reading

Key Exclusion Criteria:

* Known infiltrative or storage disorder causing cardiac hypertrophy that mimics oHCM, such as Fabry disease, amyloidosis, or Noonan syndrome with LV hypertrophy
* History of syncope or sustained ventricular tachyarrhythmia with exercise within 6 months prior to Screening
* History of resuscitated sudden cardiac arrest (at any time) or known history of appropriate implantable cardioverter defibrillator (ICD) discharge for life-threatening ventricular arrhythmia within 6 months prior to Screening
* Paroxysmal, intermittent atrial fibrillation with atrial fibrillation present at Screening
* Persistent or permanent atrial fibrillation not on anticoagulation for at least 4 weeks prior to Screening and/or not adequately rate controlled within 6 months prior to Screening
* Treatment (within 14 days prior to Screening) or planned treatment during the study with disopyramide or ranolazine
* Treatment (within 14 days prior to Screening) or planned treatment during the study with a combination of β-blockers and calcium channel blockers
* LVOT gradient with Valsalva maneuver <30 mmHg at Screening
* Has been successfully treated with invasive septal reduction (surgical myectomy or percutaneous alcohol septal ablation [ASA]) within 6 months prior to Screening or plans to have either of these treatments during the study
* ICD placement within 2 months prior to Screening or planned ICD placement during the study
* Has a history or evidence of any other clinically significant disorder, condition, or disease that, in the opinion of the investigator, would pose a risk to participant safety or interfere with the study evaluation, procedures, or completion
* Prior treatment with cardiotoxic agents such as doxorubicin or similar

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2018-05-29 (Actual); Primary Completion 2020-03-14 (Actual); Study Completion 2020-05-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Information Team, Study Director — MyoKardia, Inc.
Locations (71):
- United States (29):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Cedars-Sinai Medical Center (Smidt Heart Institute), Los Angeles, California
  - UCSF School of Medicine, San Francisco, California
  - Stanford University, Stanford, California
  - Yale New Haven Hospital, New Haven, Connecticut
  - Mayo Clinic Jacksonville - PPDS, Jacksonville, Florida
  - Northwestern University, Chicago, Illinois
  - University Of Iowa Hospitals And Clinics, Iowa City, Iowa
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Spectrum Health, Grand Rapids, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - NYU Langone Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Duke Cardiology at Southpoint, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - St. Luke's Cardiology Associates, Bethlehem, Pennsylvania
  - University of Pennsylvania (Penn Heart and Vascular Center), Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center Presbyterian, Pittsburgh, Pennsylvania
  - Methodist University Hospital, Memphis, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - University of Texas Houston Medical School, Houston, Texas
  - Intermountain Medical Center, Salt Lake City, Utah
  - University of Utah, Salt Lake City, Utah
  - University of Virginia Health System, Charlottesville, Virginia
  - University of Washington Medical Center, Seattle, Washington
- Belgium (3):
  - UZ Antwerpen, Edegem, Antwerpen
  - Onze-Lieve-Vrouwziekenhuis, Aalst, Oost-Vlaanderen
  - Hôpital Erasme, Brussels
- Czechia (2):
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Institut Klinicke a Experimentalni Mediciny, Prague
- Denmark (3):
  - Aarhus Universitetshospital, Aarhus N
  - Bispebjerg Hospital, København NV
  - Odense Universitetshospital, Odense
- France (4):
  - CHRU Nantes, Nantes, Loire-Atlantique
  - Groupe Hospitalier Pitié Salpétrière, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpital de Rangueil, Toulouse
- Germany (7):
  - University Medicine Göttingen, Göttingen, Neidersachsen
  - Kerckhoff-Klinik-Forschungs-GmbH, Bad Nauheim
  - Charité Campus Buch - Experimental and Clinical Research Center, Berlin
  - Charité - Universitätsmedizin Berlin, Berlin
  - Cardiologicum Dresden und Pirna, Dresden
  - University Clinic Heidelberg - PPDS, Heidelberg
  - Universitatsklinikum Schleswig-Holstein, Kiel
- Israel (7):
  - Tel Aviv Sourasky Medical Center, Tel Aviv, Tel Aviv
  - Barzilai Medical Center, Ashkelon
  - Hadassah Medical Center PPDS -, Jerusalem
  - Rabin Medical Center - PPDS, Petah Tikva
  - The Chaim Sheba Medical Center - The Edmond and Lily Safra Children's Hospital, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - ZIV Medical Center, Safed
- Azienda Ospedaliera Universitaria Careggi, Florence, Italy
- Netherlands (2):
  - Maastricht University Medical Center, Maastricht, Limburg
  - Erasmus MC, Rotterdam, South Holland
- Poland (4):
  - Collegium Medicum Uniwersytetu Jagiellonskiego, Krakow, Lesser Poland Voivodeship
  - Kardio Klinika Brynów, Katowice, Silesian Voivodeship
  - Szpital Kliniczny Przemienienia Panskiego Uniwesytetu Medycznego im. Karola Marcinkowskiego, Poznan
  - Instytut Kardiologii im Prymasa Tysiaclecia Kardynala Stefana Wyszynskiego, Warsaw
- Portugal (2):
  - Hospital Garcia de Orta, Almada
  - Hospital da Luz, Lisbon
- Spain (5):
  - Hospital Universitario Virgen de La Arrixaca, El Palmar, Murcia
  - Hospital Universitario A Coruña, A Coruña
  - Hospital Universitario Puerta de Hierro - Majadahonda, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario Virgen Macarena, Seville
- United Kingdom (2):
  - University Hospital of Wales, Cardiff, South Glamergon
  - St Bartholomew's Hospital, London

REFERENCES:
- [Derived] Wang A, Lakdawala NK, Abraham TP, Nilles EK, Wojdyla DM, Owens AT, Bach RG, Saberi S, Sehnert A, Cresci S. Association Between age or Duration of Diagnosis in Obstructive Hypertrophic Cardiomyopathy and Response to Mavacamten Treatment: Exploratory Analysis of the EXPLORER-HCM Trial. J Card Fail. 2025 Jun;31(6):901-911. doi: 10.1016/j.cardfail.2024.10.449. Epub 2024 Dec 7. PMID 39653325
- [Derived] Arnold SV, Gosch KL, Dolan C, Fine JT, Masri A, Saberi S, Wang A, Elliott PM, Hegde SM, Lam J, Sehnert AJ, Cresci S, Bach RG, Spertus JA. Association of Echocardiographic Parameters and Health Status in Patients With Obstructive Hypertrophic Cardiomyopathy: Insights From EXPLORER-HCM. Circulation. 2024 Nov 5;150(19):1560-1562. doi: 10.1161/CIRCULATIONAHA.123.067470. Epub 2024 Nov 4. No abstract available. PMID 39495835
- [Derived] Garcia-Pavia P, Oreziak A, Masri A, Barriales-Villa R, Abraham TP, Owens AT, Jensen MK, Wojakowski W, Seidler T, Hagege A, Lakdawala NK, Wang A, Wheeler MT, Choudhury L, Balaratnam G, Shah A, Fox S, Hegde SM, Olivotto I. Long-term effect of mavacamten in obstructive hypertrophic cardiomyopathy. Eur Heart J. 2024 Dec 16;45(47):5071-5083. doi: 10.1093/eurheartj/ehae579. PMID 39217450
- [Derived] Cresci S, Bach RG, Saberi S, Owens AT, Spertus JA, Hegde SM, Lakdawala NK, Nilles EK, Wojdyla DM, Sehnert AJ, Wang A. Effect of Mavacamten in Women Compared With Men With Obstructive Hypertrophic Cardiomyopathy: Insights From EXPLORER-HCM. Circulation. 2024 Feb 13;149(7):498-509. doi: 10.1161/CIRCULATIONAHA.123.065600. Epub 2023 Nov 14. PMID 37961906
- [Derived] Wang A, Spertus JA, Wojdyla DM, Abraham TP, Nilles EK, Owens AT, Saberi S, Cresci S, Sehnert A, Lakdawala NK. Mavacamten for Obstructive Hypertrophic Cardiomyopathy With or Without Hypertension: Post-Hoc Analysis of the EXPLORER-HCM Trial. JACC Heart Fail. 2024 Mar;12(3):567-579. doi: 10.1016/j.jchf.2023.07.030. Epub 2023 Oct 18. PMID 37855754
- [Derived] Wheeler MT, Olivotto I, Elliott PM, Saberi S, Owens AT, Maurer MS, Masri A, Sehnert AJ, Edelberg JM, Chen YM, Florea V, Malhotra R, Wang A, Oreziak A, Myers J. Effects of Mavacamten on Measures of Cardiopulmonary Exercise Testing Beyond Peak Oxygen Consumption: A Secondary Analysis of the EXPLORER-HCM Randomized Trial. JAMA Cardiol. 2023 Mar 1;8(3):240-247. doi: 10.1001/jamacardio.2022.5099. PMID 36652223
- [Derived] Nassif M, Fine JT, Dolan C, Reaney M, Addepalli P, Allen VD, Sehnert AJ, Gosch K, Spertus JA. Validation of the Kansas City Cardiomyopathy Questionnaire in Symptomatic Obstructive Hypertrophic Cardiomyopathy. JACC Heart Fail. 2022 Aug;10(8):531-539. doi: 10.1016/j.jchf.2022.03.002. Epub 2022 May 4. PMID 35902155
- [Derived] Reaney M, Addepalli P, Allen V, Spertus JA, Dolan C, Sehnert AJ, Fine JT. Longitudinal Psychometric Analysis of the Hypertrophic Cardiomyopathy Symptom Questionnaire (HCMSQ) Using Outcomes from the Phase III EXPLORER-HCM Trial. Pharmacoecon Open. 2022 Jul;6(4):575-586. doi: 10.1007/s41669-022-00340-8. Epub 2022 Jun 20. PMID 35718845
- [Derived] Hegde SM, Lester SJ, Solomon SD, Michels M, Elliott PM, Nagueh SF, Choudhury L, Zemanek D, Zwas DR, Jacoby D, Wang A, Ho CY, Li W, Sehnert AJ, Olivotto I, Abraham TP. Effect of Mavacamten on Echocardiographic Features in Symptomatic Patients With Obstructive Hypertrophic Cardiomyopathy. J Am Coll Cardiol. 2021 Dec 21;78(25):2518-2532. doi: 10.1016/j.jacc.2021.09.1381. PMID 34915982
- [Derived] Xie J, Wang Y, Xu Y, Fine JT, Lam J, Garrison LP. Assessing health-related quality-of-life in patients with symptomatic obstructive hypertrophic cardiomyopathy: EQ-5D-based utilities in the EXPLORER-HCM trial. J Med Econ. 2022 Jan-Dec;25(1):51-58. doi: 10.1080/13696998.2021.2011301. PMID 34907813
- [Derived] Burstein Waldman C, Owens A. A plain language summary of the EXPLORER-HCM study: mavacamten for obstructive hypertrophic cardiomyopathy. Future Cardiol. 2021 Oct;17(7):1269-1275. doi: 10.2217/fca-2021-0044. Epub 2021 May 21. PMID 34018809
- [Derived] Spertus JA, Fine JT, Elliott P, Ho CY, Olivotto I, Saberi S, Li W, Dolan C, Reaney M, Sehnert AJ, Jacoby D. Mavacamten for treatment of symptomatic obstructive hypertrophic cardiomyopathy (EXPLORER-HCM): health status analysis of a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet. 2021 Jun 26;397(10293):2467-2475. doi: 10.1016/S0140-6736(21)00763-7. Epub 2021 May 15. PMID 34004177
- [Derived] Olivotto I, Oreziak A, Barriales-Villa R, Abraham TP, Masri A, Garcia-Pavia P, Saberi S, Lakdawala NK, Wheeler MT, Owens A, Kubanek M, Wojakowski W, Jensen MK, Gimeno-Blanes J, Afshar K, Myers J, Hegde SM, Solomon SD, Sehnert AJ, Zhang D, Li W, Bhattacharya M, Edelberg JM, Waldman CB, Lester SJ, Wang A, Ho CY, Jacoby D; EXPLORER-HCM study investigators. Mavacamten for treatment of symptomatic obstructive hypertrophic cardiomyopathy (EXPLORER-HCM): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet. 2020 Sep 12;396(10253):759-769. doi: 10.1016/S0140-6736(20)31792-X. Epub 2020 Aug 29. PMID 32871100
- [Derived] Ho CY, Olivotto I, Jacoby D, Lester SJ, Roe M, Wang A, Waldman CB, Zhang D, Sehnert AJ, Heitner SB. Study Design and Rationale of EXPLORER-HCM: Evaluation of Mavacamten in Adults With Symptomatic Obstructive Hypertrophic Cardiomyopathy. Circ Heart Fail. 2020 Jun;13(6):e006853. doi: 10.1161/CIRCHEARTFAILURE.120.006853. Epub 2020 Jun 5. PMID 32498620

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects who met all of the inclusion criteria and none of the exclusion criteria were enrolled into the study and were randomized 1:1 to receive mavacamten (2.5, 5, 10, or 15 mg capsule) or placebo once daily for 30 weeks, followed by an 8 week post-treatment period. In total, 429 participants were assessed for eligibility and 251 were enrolled from 68 sites in the United States and EMEA.
Groups:
- Mavacamten (MYK-461): Mavacamten: mavacamten capsules
  One mavacamten 2.5, 5, 10, or 15 mg capsule once daily by mouth for 30 weeks. The starting dose of mavacamten was 5 mg once daily by mouth. At Week 8 and Week 14, mavacamten dose may have been up-titrated for individual subjects based on prespecified criteria. Down-titration was possible at Week 6, Week 8, Week 14, Week 18, Week 22 and Week 26 for individual subjects based on prespecified criteria.
- Placebo: Placebo: placebo capsule
  One placebo-to-match mavacamten capsule once daily by mouth for 30 weeks. A universal placebo capsule to match all strengths of mavacamten had the same appearance as mavacamten capsules but did not include the active ingredient.
Period: Overall Study
Arm/Group | Mavacamten (MYK-461) | Placebo
Started | 123 | 128
Completed | 119 | 125
Not Completed | 4 | 3
Not completed — Death | 0 | 1
Not completed — Did not complete Week 30 assessments due to scheduling conflict | 1 | 0
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Week 30 not completed due to circumstances surrounding the COVID-19 pandemic | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mavacamten (MYK-461) | Placebo | Total
Number analyzed (Participants) | 123 | 128 | 251
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 78 | 88 | 166
  >=65 years | 45 | 40 | 85
Age, Continuous [Median (Full Range); unit: years] | 60 [26 to 82] | 60 [18 to 81] | 60 [18 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 45 | 102
  Male | 66 | 83 | 149
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 4 | 12
  Not Hispanic or Latino | 114 | 119 | 233
  Unknown or Not Reported | 1 | 5 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 5 | 6
  White | 115 | 114 | 229
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 6 | 9

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving A Clinical Response
Description: A positive clinical response (value="YES") is defined as having achieved either an improvement of at least 1.5 mL/kg/min in peak oxygen consumption (pVO2) as determined by cardiopulmonary exercise testing (CPET) and a reduction of one or more class in New York Heart Association (NYHA) functional classification (e.g.I, II, III, or IV) -OR- an improvement of 3.0 mL/kg/min or more in pVO2 with no worsening in NYHA Functional Class.
Time Frame: 30 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Mavacamten (MYK-461): Mavacamten: mavacamten capsules
  One mavacamten 2.5, 5, 10, or 15 mg capsule once daily by mouth for 30 weeks. The starting dose of mavacamten was 5 mg once daily by mouth. At Week 6, Week 8, and Week 14, mavacamten dose may have been up-titrated or down-titrated for individual subjects based on prespecified criteria.
Arm/Group | Mavacamten (MYK-461) | Placebo
Number analyzed (Participants) | 123 | 128
Participants | 45 | 22

2. Secondary Outcome: Changes From Baseline to Week 30 in Post Exercise in LVOT Peak Gradient.
Description: The post-exercise LVOT gradient was measured from echocardiograms obtained at baseline and week 30 following a study-specified exercise protocol and read by the Cardiovascular Imaging Core Laboratory (CICL, Boston MA). Change from baseline was determined as per the study statistical analysis plan and compared between treatment arms.
Time Frame: 30 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Mavacamten (MYK-461) | Placebo
Number analyzed (Participants) | 117 | 122
mmHg | -47 (40.3) | -10 (29.6)

3. Secondary Outcome: Change From Baseline to Week 30 in pVO2 as Assessed by CPET
Description: Cardiopulmonary exercise testing (CPET) was performed at baseline and week 30 following a study-specified protocol and peak oxygen consumption (pVO2) was determined by the Cardiovascular Metabolic Disease Research Institute (CMDRI, Palo Alto, CA). Change from baseline was determined as per the study statistical analysis plan and compared between treatment arms.
Time Frame: 30 weeks
Measure: Mean (Standard Deviation); unit: mL/kg/min
Arm/Group | Mavacamten (MYK-461) | Placebo
Number analyzed (Participants) | 120 | 125
mL/kg/min | 1.4 (3.12) | -0.05 (3.02)

4. Secondary Outcome: Proportion of Participants With at Least 1 Class Improvement in NYHA Functional Class From Baseline to Week 30
Description: New York Heart Association (NYHA) functional classification was determined by the principal investigator at baseline and at specified timepoints in the study. At baseline, all subjects were NYHA Class II or III. For the secondary outcome, NYHA class at Week 30 was compared to baseline and the proportion of subjects with an improvement of at least one class was determined, and the difference between treatment groups was analyzed. The proportion was also multiplied by 100 to provide the result as a percent.
Time Frame: 30 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Mavacamten (MYK-461) | Placebo
Number analyzed (Participants) | 123 | 128
Participants | 80 | 40

5. Secondary Outcome: Change From Baseline to Week 30 in Participant-reported Health-related Quality of Life as Assessed by the KCCQ Score
Description: The Kansas City Cardiomyopathy Questionnaire (KCCQ) is a patient reported outcome instrument with minimum score = 0 and maximum score = 100 where higher score indicates better health status. There are no units to the score. The instrument utilizes a recall period of 2 weeks over which patients describe the frequency and severity of their symptoms, their physical and social limitations, and how they perceive their heart failure symptoms to affect their quality of life. The KCCQ clinical summary (KCCQ-CS) score, a prespecified secondary outcome of EXPLORER-HCM, combines the physical limitation and total symptom scores.
Time Frame: 30 weeks
Measure: Mean (Standard Deviation); unit: Scores on Scale
Arm/Group | Mavacamten (MYK-461) | Placebo
Number analyzed (Participants) | 92 | 88
Scores on Scale | 13.6 (14.42) | 4.2 (13.68)

6. Secondary Outcome: Change From Baseline to Week 30 in Participant-reported Severity of HCM Symptoms as Assessed by the HCMSQ Score
Description: The Hypertrophic Cardiomyopathy Symptom Questionnaire (HCMSQ) is a patient reported outcome instrument that is a daily self-administered 11-item questionnaire. The HCMSQ assesses the core symptoms of HCM (tiredness/fatigue, heart palpitations, chest pain, dizziness, and shortness of breath). The Shortness of Breath domain score, a pre-specified secondary outcome of EXPLORER-HCM, assesses the frequency and severity of shortness of breath. The minimum score = 0 and maximum score = 18 where lower score indicates better health status. There are no units to the score.
Time Frame: 30 weeks
Measure: Mean (Standard Deviation); unit: Scores on Scale
Arm/Group | Mavacamten (MYK-461) | Placebo
Number analyzed (Participants) | 85 | 86
Scores on Scale | -2.8 (2.68) | -0.9 (2.41)

ADVERSE EVENTS:
Time Frame: Treatment-Emergent Adverse Events (TEAEs) were summarized for the on-treatment period (Day 1 to Week 30) and for the treatment-emergent period (Day 1 to Week 38).
Description: Treatment with mavacamten was well tolerated with an overall completion rate > 97%, with a balanced AE profile between treatment arms through 30 weeks of treatment. It is notable that the TEAE rate did not increase in the mavacamten group with 8 weeks of additional observation during study drug washout. Adverse event data included below is through Week 38.
Groups:
- Placebo: Placebo: placebo oral capsule
  One placebo-to-match mavacamten capsule once daily by mouth for 30 weeks. A universal placebo capsule to match all strengths of mavacamten had the same appearance as mavacamten capsules but did not include the active ingredient. Placebo dose to match mavacamten capsule was administered once daily by mouth.
Arm/Group | Mavacamten (MYK-461) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/123 | 1/128
Serious Adverse Events (participants affected / at risk) | 14/123 | 12/128
Other Adverse Events (participants affected / at risk) | 108/123 | 104/128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mavacamten (MYK-461) (N=123) | Placebo (N=128)
Atrial Fibrillation (Cardiac disorders) | 3 | 5
Stress cardiomyopathy (Cardiac disorders) | 2 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 1
Cardiac Failure (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Cardiogenic shock (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Systolic dysfunction (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Atrial septal defect (Congenital, familial and genetic disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 0
Sudden Death (General disorders) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 2
Bacterial colitis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Forearm Fracture (Injury, poisoning and procedural complications) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
SLE (Musculoskeletal and connective tissue disorders) | 1 | 0
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Syncope (Nervous system disorders) | 3 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Device inappropriate shock delivery (Product Issues) | 1 | 0
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mavacamten (MYK-461) (N=123) | Placebo (N=128)
Atrial Fibrillation (Cardiac disorders) | 10 | 10
Palpitations (Cardiac disorders) | 7 | 10
Angina pectoris (Cardiac disorders) | 3 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 18 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 4
Dizziness (Nervous system disorders) | 26 | 17
Headache (Nervous system disorders) | 15 | 10
Syncope (Nervous system disorders) | 7 | 2
Fatigue (General disorders) | 7 | 7
Diarrhoea (Gastrointestinal disorders) | 5 | 7
Gastroesophageal reflux disease (Gastrointestinal disorders) | 7 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 2
Nasopharyngitis (Infections and infestations) | 15 | 19
Upper respiratory tract infection (Infections and infestations) | 10 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2019-10-04): https://cdn.clinicaltrials.gov/large-docs/45/NCT03470545/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-21): https://cdn.clinicaltrials.gov/large-docs/45/NCT03470545/SAP_001.pdf